CLINICAL TRIAL: NCT01500798
Title: A Pharmacodynamic Study of Measured Glomerular Filtration Rate Assessed by Tc99m-DTPA in Patients With Chronic Kidney Disease and Type 2 Diabetes
Brief Title: A Pharmacodynamic Study of Measured Glomerular Filtration Rate in Patients With Chronic Kidney Disease and Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IDMC recommendation for safety concerns
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-1005
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Bardoxolone methyl (Experimental)
  Interventions: Drug: 20 mg bardoxolone methyl

INTERVENTIONS:
Drug: 20 mg bardoxolone methyl — 20 mg, oral, once daily
  Arms: Bardoxolone methyl
Drug: Placebo — Oral, once daily
  Arms: Placebo

SUMMARY:
This is a 24-week multi-center, double-blind, randomized, exploratory study of bardoxolone methyl treatment in 18 patients with Stage 3 CKD (eGFR greater than or equal to 30.0 to less than 60.0 ml/min/1.73m2) and diabetes to ensure at least 15 patients complete the study for evaluation of the primary endpoints.

DETAILED DESCRIPTION:
This study was previously posted by Reata Pharmaceuticals. In September 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Screening eGFR ≥ 30.0 and < 60.0 mL/min/1.73 m2;
* A history of type 2 diabetes; diagnosis should have been made at ≥ 30 years of age (if diabetes developed at a younger age, a fasting C-peptide level must be ≥ 0.1 ng/mL to confirm type 2 diabetes);
* Male or female patients at least 18 years of age;
* Treatment with an angiotensin converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB) for at least 6 weeks prior to Screening Visit and during screening. The dosage of ACE inhibitor and/or ARB must be stable for 2 weeks prior to Screening Visit A and during screening (i.e., no change in dosage or medication). Patients not taking an ACE inhibitor and/or ARB, or taking an ACE inhibitor and/or ARB at levels below the goal dose set by K/DOQI guidelines (See Appendix 3) should have a documented medical contraindication (e.g., hyperkalemia, dry cough, angioedema), which the investigator must discuss with the appropriate medical monitor;
* Albumin/creatinine ratio (ACR) < 300 mg/g;
* Mean systolic blood pressure (SBP) must be ≤ 160 mmHg and ≥ 105 mmHg and mean diastolic blood pressure (DBP) must be < 90 mmHg during screening; both mean SBP and mean DBP (determined as the average of three readings) must be within the described range;
* Willing to practice methods of birth control (both males who have partners of childbearing potential and females of childbearing potential, [see Section 9.7]) during screening, while taking study drug and for at least 30 days after the last dose of study drug is ingested;
* Willing and able to cooperate with all aspects of the protocol;
* Willing and able to give written informed consent for study participation and provide consent for access to medical data according to appropriate local data protection legislation, allowing authorization to access medical records that describe events captured in the endpoints.

Exclusion Criteria:

* Type 1 diabetes mellitus (juvenile onset). If a history of diabetic ketoacidosis exists, a C-peptide level must confirm type 2 diabetes;
* Known non-diabetic renal disease (e.g., known polycystic kidney disease or family history of a hereditary form of kidney disease) [nephrosclerosis superimposed on diabetic kidney disease is acceptable];
* Ongoing clinical investigation with evidence (e.g., unexplained hematuria or red blood cell or white blood cell casts) suggesting non-diabetic renal disease other than nephrosclerosis;
* History of a renal donation, transplant or a planned transplant from a living donor during the study;
* Hemoglobin A1c level > 9.0% (75 mmol/mol) during screening;
* Acute dialysis or acute kidney injury within 12 weeks prior to screening or during screening;
* Clinical signs and/or symptoms of uremia and expected need for renal replacement therapy within 12 weeks following randomization, as assessed by the investigator;
* Recently active cardiovascular disease defined as:

  * Unstable angina pectoris within 12 weeks before study randomization;
  * Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 12 weeks before study randomization;
  * Cerebrovascular accident, including transient ischemic attack within 12 weeks before study randomization;
  * Current diagnosis of Class III or IV NYHA congestive heart failure (Appendix 4);
* Clinical diagnosis of severe obstructive valvular heart disease or severe obstructive hypertrophic cardiomyopathy;
* Atrioventricular block, 2o or 3o, not successfully treated with a pacemaker;
* Diagnostic or interventional procedure that required a contrast agent within 30 days prior to baseline mGFR visit 1 or planned during the study;
* Systemic immunosuppression for more than 2 weeks, cumulatively, within the 12 weeks prior to randomization or anticipated need for immunosuppression during the study;
* Total bilirubin, aspartate transaminase (AST), or alanine transaminase (ALT) level greater than the upper limit of normal (ULN) or alkaline phosphatase level greater than two times the ULN on ANY screening laboratory test result;
* Female patients who are pregnant, intend to become pregnant during the study, or are nursing;
* BMI < 18.5 kg/m2;
* Known hypersensitivity to any component of the study drug;
* Current history of drug or alcohol abuse, as assessed by the investigator;
* Clinically significant infection requiring intravenous administration of antibiotics or hospitalization within 6 weeks prior to Screening Visit or during screening;
* Diagnosis or treatment of a malignancy in the past 5 years, excluding non-melanoma skin cancer and carcinoma in situ of the cervix;
* A clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the patient while involved in the study;
* Unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function;
* Participation in a clinical study involving any intervention within 30 days prior to randomization, concurrent participation in such a study, or participation in a prior clinical study involving bardoxolone methyl in any form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2013-10-01 (Actual)

PRIMARY OUTCOMES:
Measured GFR assessed by plasma clearance of Tc99m-DTPA | 24 weeks
  Measured GFR assessed by plasma clearance of Tc99m-DTPA at Baseline mGFR assessment 1, Baseline mGFR assessment 2, and at Weeks 8, 16 and 20

SECONDARY OUTCOMES:
Measured GFR assessed by gama camera assessment of renal uptake of Tc99m-DTPA | 24 weeks
  Measured GFR assessed by gama camera assessment of renal uptake of Tc99m-DTPA at Baseline mGFR assessment 1, Baseline mGFR assessment 2, and at Weeks 8, 16 and 20
Circulating endothelial cell assessments | 24 weeks
  Circulating endothelial cell assessments at Baseline mGFR assessment 1 and at Weeks 8 and 20

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/